CLINICAL TRIAL: NCT07126899
Title: Hand Tendon Injuries: Investigation of Attention Deficit, Hyperactivity, Impulsivity, Anger, and Anxiety Levels - Case-Control Study
Brief Title: Hand Tendon Injuries: An Investigation Of Attention Deficit Disorder
Acronym: Tendon-ADHD
Status: Active, not recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-GOKAEK-2411_2024.10.16_16
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; Tendon Injuries
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Tendon Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tendon injuries cause significant disability, loss of work capacity, and economic burden. The injury itself and its consequences impact individuals not only in terms of their ability to work but also socially and psychologically. Identifying the characteristics of these injuries, many of which occur through preventable mechanisms, is crucial for guiding preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Those with tendon injuries,
* Those aged between 18 and 65,
* Those with good cognitive function,

Exclusion Criteria:

* Tendon injury diagnosis is uncertain,
* Cognitive function is poor,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The medical history and results of completed scales for patients aged between 18 and 65 with good cognitive function will be recorded on the patient form. The medical history and results of completed scales for healthy individuals aged between 18 and 65 with good cognitive function, who are of similar age and gender to the patient group, have no tendon injuries, and will be recorded on the control form.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
ASRS-Barratt-Anger | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University, Yozgat, Turkey (Türkiye)